CLINICAL TRIAL: NCT00883272
Title: Assessment of Femarelle (DT56a), a Novel SERM, Effect on the Clotting Time in Normal and Thrombophililic Postmenopausal Women
Brief Title: Effect of DT56a (Femarelle) on the Coagulation System in the Treatment of Postmenopausal Women
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 03-0670-0
Record Dates: First submitted 2009-04-16; First posted 2009-04-17 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Menopause; Thrombophilia
Keywords: Menopause; Thrombophilia; factor V Leiden; Estrogen Replacement Therapy; Hypercoagulability; Venous Thrombosis
MeSH Terms: conditions — Thrombophilia; Venous Thrombosis | interventions — DT56a

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples were collected in evacuated tubes (Vacutainer, Becton Dickinson) at baseline, eight weeks, and one year.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal Controls: 25 women with CADP-CT > 66 seconds were treated with Femarelle
  Interventions: Dietary Supplement: DT56a (Femarelle) [Se-cure pharmaceuticals, Dalton, Israel]
- Thrombophilic: Seven women in cohort of a previous study were found to have shortened closure times (CADP-CT < 61s) at time of enrollment. They all underwent genetic testing for a hypercoagulable state.
  Interventions: Dietary Supplement: DT56a (Femarelle) [Se-cure pharmaceuticals, Dalton, Israel]

INTERVENTIONS:
Dietary Supplement: DT56a (Femarelle) [Se-cure pharmaceuticals, Dalton, Israel] — a unique enzymatic isolate of the active complex in Tofu

SUMMARY:
The purpose of this study is to determine if Femeralle (DT56a) has an effect on the coagulation system, measured by platelet adhesion and aggregation, of normal and thrombophilic postmenopausal women.

DETAILED DESCRIPTION:
Women using hormone therapy (HT) are at an increased relative risk of venous thromboembolism (VTE). The frequency of inherited Factor V Leiden and other risk factors for VTE in the general population is estimated at 5-10%. This population has a 5-21 fold greater risk to develop VTE. Therefore, given the high thrombotic risk for the combination of hormone use and hereditary prothrombotic abnormalities these women's symptoms frequently go untreated for lack of alternative therapies. DT56a (Femarelle) is a soy derived compound that has been shown to act as a novel selective estrogen receptor modulator (SERM) in the alleviation of menopausal symptoms and prevention of postmenopausal bone loss without effecting the endometrium or the sex hormone blood profile. The research question of the current study is to assess the effect of femeralle on the coagulation system and determine if it is a reasonable and safe alternative for the treatment of menopausal symptoms in thrombophilic women.

ELIGIBILITY:
Inclusion Criteria:

* No previous exogenous estrogen exposure
* Symptomatic Menopause: hot flashes, sleep disturbance, or other symptoms related to estrogen deficiency
* Menopausal (see above)

Exclusion Criteria:

* History of bleeding or thrombotic disorder
* History of malignancy (particularly Breast Cancer)
* Diabetics
* Coronary Artery Disease
* Liver Disease
* Concurrent Anticoagulation therapy

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Peri- and postmenopausal women aged 40-67. Menopause defined as a FSH > 40 and no menses for > 1 year.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-01; Primary Completion 2009-01 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The PFA-100 (Dade Behring, Inc.) device was used to evaluate platelet adhesion and aggregation. Clotting time (sec.) was recorded and defined as the time for blood to block a collagen membrane coated with epinephrine (CEPI) or ADP (CADP). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lila Nachtigall, MD, Principal Investigator — NYU Langone Health
Locations (1):
- 251 East 33rd Street, New York, New York, United States

REFERENCES:
- [Background] Flaumenhaft R, Nachtigall M, Lowenstein J, Nachtigall L, Nachtigall R, Nachtigall L. Association of oral but not transdermal estrogen therapy with enhanced platelet reactivity in a subset of postmenopausal women. Menopause. 2009 Mar-Apr;16(2):407-12. doi: 10.1097/gme.0b013e3181833886. PMID 18989235
- [Background] Somjen D, Katzburg S, Knoll E, Hendel D, Stern N, Kaye AM, Yoles I. DT56a (Femarelle): a natural selective estrogen receptor modulator (SERM). J Steroid Biochem Mol Biol. 2007 May;104(3-5):252-8. doi: 10.1016/j.jsbmb.2007.03.004. Epub 2007 Mar 14. PMID 17428655